CLINICAL TRIAL: NCT00578708
Title: Closure of Perimembranous Ventricular Septal Defects With The AMPLATZER® Membranous VSD OCCLUDER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AGA-008; G020202
Record Dates: First submitted 2007-12-20; First posted 2007-12-21 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-02

CONDITIONS: Membranous Ventricular Septal Defects
Keywords: membranous; ventricular; septal; defect; VSD

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Device: AMPLATZER Membranous VSD Occluder

INTERVENTIONS:
Device: AMPLATZER Membranous VSD Occluder — Device closure with the AMPLATZER Membranous VSD Occluder

SUMMARY:
The purpose of this feasibility study is to investigate the safety of the AMPLATZER® Membranous VSD Occluder for the treatment of hemodynamically significant Perimembranous Ventricular Septal Defects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hemodynamically significant Perimembranous ventricular septal defects

Exclusion Criteria:

* Patients < 8 kg
* Supracristal ventricular septal defects
* Left ventricle to right atrium shunting
* Prolapse of the aortic valve
* Right to left shunting through the defect
* Perimembranous VSD with an aneurysm and multiple shunts which can not be successfully closed with one device
* Patients with <2mm aortic rim
* Sepsis (local/generalized)
* Complex heart lesions such as atrioventricular canal defect or Tetralogy of Fallot.
* Patients who are ASA intolerant
* Unable to be followed for the duration of the clinical trial
* Inability to obtain informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2003-09; Primary Completion 2010-03 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Closure of perimembranous Ventricular Septal Defects | 5 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University Medical Center, St Louis, Missouri
  - Children's Hospital UN/CU), Omaha, Nebraska
  - Columbia University, New York, New York
  - Columbus Children's Hospital, Columbus, Ohio
  - Medical University of South Carolina, Charleston, South Carolina